CLINICAL TRIAL: NCT00000923
Title: Treatment Rollover for Subjects Formerly on ACTG 328 With Subcutaneous Interleukin-2 (IL-2) in Combination With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Treatment With Interleukin-2 (IL-2) Plus Combination Anti-HIV-Drug Therapy (HAART) for Patients Formerly in ACTG 328
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5051; 10205 (Registry Identifier: DAIDS ES Registry Number); Substudy ACTG A5052s; Substudy ACTG A5053s; Substudy ACTG A5054s; Substudy ACTG A5094s; AACTG A5051; ACTG A5051
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Drug Therapy, Combination; CD4 Lymphocyte Count; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine; Didanosine; aldesleukin

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine
Drug: Aldesleukin

SUMMARY:
This study examines the long-term effects of interleukin-2 (IL-2) in combination with anti-HIV drugs, or highly active antiretroviral therapy (HAART). The purpose of this study is to see if IL-2 can increase the number of CD4 cells (cells of the immune system which fight infection) in HIV-infected patients who have completed ACTG 328.

HAART is often successful in decreasing viral load (level of HIV in the blood), but these drugs have not been able to restore the immune systems of HIV-infected patients. IL-2 is a substance naturally produced by the body's immune cells. In ACTG 328, IL-2 is tested to see if it can increase the number of CD4 cells and "boost" a patient's immune system. This study is a follow-up to ACTG 328 so that patients who are benefiting from IL-2 can continue to take it and patients in the control group who do not receive IL-2 can start taking it.

DETAILED DESCRIPTION:
HIV disease is characterized by a progressive decline in CD4 cells and an increase in viral burden. Although antiretroviral therapy has been successful in controlling viral levels, its effects on CD4 cell counts have been modest. Intermittently administered IL-2 in the presence of HAART has been shown to increase CD4 cell counts, decrease lymphocyte activation markers, and increase certain lymphocyte functional activity in patients with early-stage HIV infection. ACTG 328 evaluated the effects of intravenous and/or subcutaneously administered IL-2 in conjunction with HAART in a group of more advanced HIV-infected patients over an 18- to 22-month period. As patients were enrolled in this study over an 18-month period, a follow-up protocol is required to provide continued IL-2 therapy for patients responding to IL-2 and patients in the control group who wish to receive this drug.

This study enrolls patients who participated in ACTG 328. Patients in Arm I of ACTG 328 (the control group receiving HAART only) who have a viral load of 5,000 copies/ml or less register for Step II. Patients in Step II receive subcutaneous [SC] IL-2 in combination with HAART. IL-2 is administered for 5 days every 8 weeks for the first 3 cycles. For subsequent cycles, the interval between cycles may be extended in 8-week increments for a maximum of 24 weeks, provided the patient's bimonthly CD4 count exceeds 500 cells/mm3. Patients in Arm I who have a viral load greater than 5,000 copies/ml register for Step I which requires a change in antiretroviral therapy. Patients who then achieve viral levels of 5,000 copies/ml or less may begin to receive IL-2 no earlier than 4 weeks and no later than 12 weeks after the change in HAART regimen. Patients whose viral load remains above 5,000 copies/ml for 12 weeks after the change in drug regimen are discontinued from the study. Patients in Arms II or III of ACTG 328 (IL-2-containing arms) who have had a 25 percent or greater increase in CD4 cell count above their Week 11 value and have a viral load of 5,000 copies/ml or less continue on SC IL-2 and HAART. Patients who meet the CD4 criteria but whose viral load is above 5,000 copies/ml change their HAART regimen. After a minimum of 4 weeks and a maximum of 12 weeks, these patients may receive IL-2 provided they have a viral load of 5,000 copies/ml or less. For this study, HAART is defined as one protease inhibitor and two nucleoside analogues. [AS PER AMENDMENT 9/16/99: All patients must receive a protease inhibitor or, with permission of the chair, a nonnucleoside reverse transcriptase inhibitor (NNRTI) plus either two nucleoside reverse transcriptase inhibitors (NRTIs) or another protease inhibitor or NNRTI.] The protease inhibitor provided on this study is indinavir (IDV). The nucleoside analogue combinations provided on this study are as follows: zidovudine (ZDV) plus didanosine (ddI), ZDV plus lamivudine (3TC), stavudine (d4T) plus 3TC, or d4T plus ddI. Other antiretroviral drugs may be used but are not provided by this study. Patients are monitored for CD4 counts at bimonthly intervals after the first IL-2 dose. CD4 counts and plasma storage for HIV RNA are done within 96 hours prior to each cycle of IL-2. Safety laboratory evaluations are obtained prior to and at the conclusion of each IL-2 course. TSH (thyroid-stimulating hormone), DTH skin testing, and real-time plasma HIV RNA are obtained at 6-month intervals.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have completed at least 84 weeks of treatment on ACTG 328.
* Have had a 25 percent or greater increase in CD4 cell count above the ACTG 328 Week 11 value (only applies to patients who received IL-2 during ACTG 328).
* Are 18 years of age or older.
* Agree to practice abstinence or use a barrier method of birth control (such as condoms) during the study. (This study has been changed. Hormonal methods of birth control such as birth control pills are no longer allowed.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have significant heart disease or are taking certain heart medications. Patients with hypertension who are being treated are eligible.
* Have taken certain medications that might affect the immune system within 4 weeks of study entry including corticosteroids, interferons, or thalidomide.
* Have taken rifampin, rifabutin, or St. John's wort within 7 days of study entry. (This study has been changed. St. John's wort was not in the original version.)
* Are taking certain investigational anti-HIV drugs.
* Are taking indinavir and any of the following within 2 weeks of study entry: cisapride, terfenadine, astemizole, midazolam, triazolam, ketoconazole, itraconazole, or delavirdine.
* Have cancer requiring chemotherapy. Local radiation therapy is allowed.
* Have untreated thyroid disease.
* Are allergic to albumin.
* Have a serious mental illness.
* Have a history of an autoimmune disease, including inflammatory bowel disease and psoriasis.
* Have a central nervous system disease or seizures, if these have been active within 1 year prior to study entry.
* Abuse drugs or alcohol.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Mitsuyasu, Study Chair; Richard Pollard, Study Chair
Locations (12):
- United States (12):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Tulane Univ. A1701 CRS, New Orleans, Louisiana
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Mt. Sinai Med. Ctr. A0404 CRS, New York, New York
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Result] Bosch RJ, Pollard RB, Landay A, Aga E, Fox L, Mitsuyasu R. Continuing or adding IL-2 in patients treated with antiretroviral therapy (ACTG Protocol A5051, a rollover trial of ACTG Protocol A328). AIDS Res Ther. 2010 Aug 5;7:30. doi: 10.1186/1742-6405-7-30. PMID 20687947